CLINICAL TRIAL: NCT01368341
Title: Tick Borne Diseases in Norwegian General Practice. A Randomized, Controlled Trial for Treatment of Erythema Migrans in Norwegian General Practice. A Comparison of Phenoxymethylpenicillin, Amoxicillin and Doxycycline.
Brief Title: Comparing 3 Antibiotic Regimes for Erythema Migrans in General Practice
Acronym: NorTick_EM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Morten Lindbaek (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Sorlandet Hospital HF (Other Government); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor-Investigator, Morten Lindbaek, Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUDRACT 2010-023747
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Erythema Migrans; Erythema Chronicum Migrans; Borreliosis; Lyme Disease; Early Lyme Disease
Keywords: Antibiotics; General Practice; Erythema migrans; Borrelia; Ticks
MeSH Terms: conditions — Glossitis, Benign Migratory; Erythema Chronicum Migrans; Borrelia Infections; Lyme Disease | interventions — Doxycycline; Penicillin V; Amoxicillin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Doxycycline (Active Comparator): Doxycycline, 100 mg, tablets, b.i.d., 14 days
  Interventions: Drug: Doxycycline
- Penicillin (Active Comparator): Phenoxymethylpenicillin tablets 650 mg. 2 tablets t.i.d. 14 days
  Interventions: Drug: Phenoxymethylpenicillin
- Amoxicillin (Active Comparator): Amoxicillin 500 mg capsula, t.i.d., 14 days
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Doxycycline — 1 tablet, 100 mg, b.i.d. 14 days
  Other Names: Doksycycline 100 mg HEXAL, no. 30
  Arms: Doxycycline
Drug: Phenoxymethylpenicillin — Tablet 650 mg, 2 tablets, t.i.d., 14 days
  Other Names: Weifapenin 650 mg, WEIFA, no. 100
  Arms: Penicillin
Drug: Amoxicillin — Capsula, 500 mg, t.i.d., 14 days
  Other Names: Amoxicillin 500 mg MYLAN, no. 30 + 20.
  Arms: Amoxicillin

SUMMARY:
Tick borne diseases are increasing in Norway. Lyme borreliosis is the most common infection. Erythema migrans is mainly diagnosed and treated in general practice. There is disagreement about what antibiotic treatment that should be given. An RCT with the three most common antibiotics used, will support data for revision of national guidelines.

DETAILED DESCRIPTION:
Comparison of phenoxymethylpenicillin, doxycycline and amoxicillin for Erythema migrans in Norwegian general practice. Every patient receives 14 days of antibiotic treatment. There are blood samples for measurement of Borrelia antibody level at day 1, 14 and 90 and questionnaires on subjective health complaints (SHC) at day 1, 90 and 360. Side symptoms and side effects are registered. For volunteers there is an additional PCR-analysis on punch biopsy from the EM for subgrouping of the Borrelia bacteria. TBE-antibodies are measured on day 14. Antibody levels and SHC-scores are compared to healthy blood donors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Erythema migrans
* Over the age of 18
* Signing an concent form after information in writing

Exclusion Criteria:

* Allergic to any of the three drugs in the study
* Under the age of 18
* Pregnancy
* Dementia or known drug abuse
* Antibiotic treatment last 14 days
* Concommitant Chemotherapy or immunomodulating therapy
* Concommitant use of medicine with potential interaction (defined in protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Duration of Erythema migrans (EM) | 1-90 days
  On day 1 duration until first the consulation is registered. Day 1-14 the EM is registered in a patient diary. On day 14 the doctor is asked whether the EM has disseapeared. If not the patient is followed by phone from the researchers. On day 90 they are additionally asked for how long it lasted.

SECONDARY OUTCOMES:
Subjective Health Complaints (SHC) | 1 year
  By questionnaire on day 1, day 90 and day 360 the patients are asked about their SHC which is a standardized set of parametres. The 3 treatment groups are compaired to each other and to 1200 healthy blood donors receiving the same questionnaire. There are 29 standardized and 3 Lyme disease related subjects to be measured.
Borrelia antibodies | 1-90 days
  Normally antibody production is not measured for EM as it is a clinical diagnosis, and less than 50 percent of EM-patients are expected to develop antibodies in the first period. However antibodies are here measured on day 1, day 14 and day 90 to see whether there are differences between the groups. Also the results will be compared to the blood donors.
Side symptoms | 1-14 days
  The EM in it self is often asymptomatic, and fever, headache and nerval palsy can be a sign of disseminated disease or co-infection. On the quiestionnaire to the pasient and doctor on day 1, in the patient diary day 1-14 and on the questionnaire to the doctor on day 14 these side symptoms are registered.
  In a potential case, where it turns out that the patient suffers from disseminated disease this will be regostered as treatment failure in the study and the patient treated and/or referred as normal.
Side effects | 1-14 days
  The antibiotic tretments are expected to be non-inferior to each other. Potensial side effects as nausea, diarrhea etc. are registered in the patients diary day 1-14 and in the doctors quiestionnaire on day 14.
Subgrouping and TBE | 1-14 days
  For volunteers there is an additional PCR-analysis on punch biopsy from the EM for subgroupring of the Borrelia bacteria. TBE-antibodies are measured on day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindbak, Professor, Principal Investigator — University of Oslo
Locations (1):
- Antibiotic Centre for Primary Care, University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Eliassen KE, Reiso H, Berild D, Lindbaek M. Comparison of phenoxymethylpenicillin, amoxicillin, and doxycycline for erythema migrans in general practice. A randomized controlled trial with a 1-year follow-up. Clin Microbiol Infect. 2018 Dec;24(12):1290-1296. doi: 10.1016/j.cmi.2018.02.028. Epub 2018 Mar 2. PMID 29505880
- See also: Information from the Antibiotic Centre for Primary Care — http://www.antibiotikasenteret.no